CLINICAL TRIAL: NCT03505177
Title: Characterization of the Gut Microbiota Composition and Activity After Three Weeks of Chitin-glucan Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathalie Delzenne (Other)
Responsible Party: Sponsor-Investigator, Nathalie Delzenne, Professor, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FiberTAG2
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Supplementation during 3 weeks with 4.5g of chitin-glucan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chitin-glucan (Experimental): Supplementation during 3 weeks with 4.5g per day of chitin-glucan fiber
  Interventions: Dietary Supplement: Chitin-glucan fiber

INTERVENTIONS:
Dietary Supplement: Chitin-glucan fiber — 4.5g per day of chitin-glucan during 3 weeks

SUMMARY:
The aim of this research study is to characterize gut microbiota composition and activity after a daily supplementation of 4.5 g of chitin-glucan during 3 weeks. For this purpose, a monocentric longitudinal intervention study without control will be performed. Fecal microbiota composition and fecal concentrations of gut microbiota-derived metabolites (bile acids, conjugated-polyunsaturated fatty acids and short-chain fatty acids) will be measured. In addition, during ten hours following the ingestion of a test meal rich in fibers, the kinetic of production of H2, methane and volatile compounds exhaled from breath will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 40 years
* Body mass index (BMI) between 18 and 25 kg/m2
* In good general health as evidenced by medical history and physical examination
* Non-smoker
* Caucasian
* H2 - producer
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Subjects presenting gastro-intestinal disorders such as ulcers, diverticulitis and inflammatory bowel diseases
* Subject presenting allergy or food intolerance (lactose, gluten,…)
* Subjects with psychiatric problems and/or using antipsychotics
* Current or recent (< 4 weeks) intake of antibiotic, probiotic, prebiotic, fiber supplement, and/or any product modulating gut transit
* Feeding particular diet such as vegetarian diet or hyper protein diet
* Chronic intake of drug, excepted contraceptive drug
* Pregnant or lactating woman or woman who did not use highly effective contraception
* Subjects who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day)
* Subjects having participated to another clinical trial two weeks before the screening test visit
* Subjects presenting an allergy or intolerance to one component of the product tested

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-22 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | Difference between day 0 and day 21
  Illumina sequencing of 16SrDNA

SECONDARY OUTCOMES:
Fecal short-chain fatty acids | Difference between day 0 and day 21
  Gas chromatography using Flame ionization detector (GC- FID)
Fecal bile acids | Difference between day 0 and day 21
  Gas chromatography-mass spectrometry (GC/MS)
Fecal conjugated-linoleic acids | Difference between day 0 and day 21
  Gas chromatography using Flame ionization detector (GC- FID)
Exhaled acetate | Difference between day 0 and day 21
  Gas chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled propionate | Difference between day 0 and day 21
  Gas chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled butyrate | Difference between day 0 and day 21
  Gas chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled C2 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled CO2 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled H2S | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled O2 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled N2 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled CH4 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled CO | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled H2 | Difference between day 0 and day 21
  Gas chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Exhaled volatile compounds | Difference between day 0 and day 21
  Gas chromatography using selected ion flow tube mass spectrometry - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - discomfort | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - nausea | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - bloating | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - flatulences | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - gastrointestinal reflux | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - cramps | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - rumbling | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - burps | 3 weeks
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - every day during the chitin-glucan supplementation
Gastro-intestinal symptom - discomfort | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - nausea | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - bloating | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - flatulences | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - gastrointestinal reflux | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - cramps | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - rumbling | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)
Gastro-intestinal symptom - burps | Difference between Day 0 and Day 21
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 10 hours following high-fiber test meal ingestion)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Investigation in Clinical Nutrition, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared by the partners from the Consortium agreement.
  * exhaled volatile metabolites
  * gut microbiota derived metabolites
  * visual analog scale data
  * concomitant medication, inclusion/exclusion criteria, adverse event, food and beverage consumption Data will be shared at the end of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study
Access Criteria: Belonging to the project Consortium